CLINICAL TRIAL: NCT03447626
Title: Post-Market Study of Robotic-Arm Assisted Unicompartmental Knee Arthroplasty in Comparison to Traditional UKA (Fixed and Mobile Bearings)
Brief Title: UKA Manual Versus UKA MAKO Robotic
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201708096
Record Dates: First submitted 2017-12-11; First posted 2018-02-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective Group- Robotic UKA Arm: Robotic UKA with the MAKO machine.
  Interventions: Device: MAKO Robotic UKA
- Control- Fixed and Mobile UKA Arm: Patients who have received fixed or mobile bearing UKA
- Control-Total Knee Arthroplasty: Patients who have had cemented or cementless total knee arthroplasty

INTERVENTIONS:
Device: MAKO Robotic UKA — Prospective UKA patient receiving unilateral knee arthroplasty using the MAKO robotic machine
  Groups: Prospective Group- Robotic UKA Arm

SUMMARY:
The purposes of this investigation is to 1) To determine if Robotic-arm assisted UKA (RA-UKA) allows for more accurate component placement than manual UKA (MI-UKA)and 2) prospectively assess the learning curve, radiographic, and clinical outcomes of use of the RIO system as it is incorporated into our clinical practice and compare it to historical data on manual UKAs and TKAs.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is known to have excellent long-term survivorship and clinical success in the management of degenerative joint disease, and remains the primary treatment for patients with bi- or tri-compartmental osteoarthritis. However, the patient population seeking knee arthroplasty is evolving, with patients being younger and more demanding on their prostheses (1). Recent investigations have highlighted that there remains a high incidence of residual symptoms including grinding/popping/clicking, swelling, and difficulties getting in and out of a car and chair, and 16% of patients remain "unsatisfied" following TKA (1).

Medial unicompartmental knee arthroplasty (UKA) remains a viable alternative to total knee arthroplasty in patients presenting with isolated, medial compartment osteoarthritis of the knee. Its use has increased in popularity in the United States, as the number of UKA performed over the last decade has increased by 30%(1). Proposed benefits of UKA include a smaller incision, less blood loss as well as shorter recovery time to functional level. Other benefits of UKAs include improved knee range of motion and better restoration of the knee kinematics (2, 5). These benefits are attributed to the less invasive nature of the procedure with preservation of the anterior and posterior cruciate ligaments, and minimal bony resections.

Unfortunately, historically the survival rate of UKA has been poor, with several reports demonstrating a survival rate of only 65-70% at 7-10 year follow-up (8, 9). These historically poor results have been attributed to instrumentation that was difficult to use, poor indications for the surgical procedure, and inadequate implant designs. More recent reports have shown 10-year survival rates ranging from 91% to 98% using both mobile-bearing and fixed-bearing UKA designs (7, 10-12). Mobile bearing UKA have a 92% survival rate at 20 years (5). However, the vast majority of these studies were performed at high-volume centers, and national joint registries have continued to demonstrate an increased rate of early failure and decreased survivorship of UKA versus TKA(13).

Recently, robotic-assisted UKA has been introduced to improve the accuracy of implant positioning (4). As implant positioning including alignment and translation in the coronal and sagittal planes and implant sizing are critical for success after UKA, the addition of robotic-assistance theoretically can improve radiographic alignment and clinical outcomes.

Currently, the most common robotic guidance system used in UKA is the Robotic Arm Interactive Orthopedic System (RIO; MAKO Surgical; Ft. Lauderdale, FLA). The purposes of this investigation is to 1) retrospectively review the radiographic and clinical outcomes of medial UKA using conventional techniques performed at our institution and 2) prospectively assess the learning curve, radiographic, and clinical outcomes of use of the RIO system as it is incorporated into our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive a robotic arm assisted UKA using the RIO navigation system will be prospectively included. All patients who have received a medial fixed or mobile UKA performed by surgeons in the Joint Preservation, Resurfacing, and Replacement Service at Washington University will be retrospectively reviewed. Also, all TKAs from a pervious study (IRB 201308057) performed by surgeons in the Joint Preservation, Resurfacing, and Replacement Service at Washington University will be retrospectively reviewed as well.

  * Patient is willing and able to comply with postoperative follow-up requirements and self-evaluations
  * Patient is willing to sign an IRB approved informed consent
  * Patient is at least 18 years of age

Exclusion Criteria:

* • Patient has a BMI < 40

  * Patient is skeletally immature
  * Patient has an active infection or suspected infection in or about the joint
  * Bone stock that is inadequate to support fixation of the prosthesis
  * Neuromuscular disorders, muscular atrophy or vascular deficiency in the affected limb rendering the procedure unjustified.
  * Patients with mental or neurological conditions which may be incapable of following instructions.
  * Blood supply limitations
  * Collateral ligament insufficiency.
  * Patients with prior HTOs or Unis.
  * Patients requiring bilateral knee arthroplasty.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unilateral arthroplasty knee patients and total Knee arthroplasty patients
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Post Op EOS measurements for alignment | 1 day- post op
  To determine if Robotic-arm assisted UKA (RA-UKA) allows for more accurate component placement than manual UKA (MI-UKA). units of measurement will be inches.

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Tsai TY, Dimitriou D, Liow MH, Rubash HE, Li G, Kwon YM. Three-Dimensional Imaging Analysis of Unicompartmental Knee Arthroplasty Evaluated in Standing Position: Component Alignment and In Vivo Articular Contact. J Arthroplasty. 2016 May;31(5):1096-101. doi: 10.1016/j.arth.2015.11.027. Epub 2015 Nov 30. PMID 26730450
- [Background] Bell SW, Anthony I, Jones B, MacLean A, Rowe P, Blyth M. Improved Accuracy of Component Positioning with Robotic-Assisted Unicompartmental Knee Arthroplasty: Data from a Prospective, Randomized Controlled Study. J Bone Joint Surg Am. 2016 Apr 20;98(8):627-35. doi: 10.2106/JBJS.15.00664. PMID 27098321
- [Background] Barrett WP, Scott RD. Revision of failed unicondylar unicompartmental knee arthroplasty. J Bone Joint Surg Am. 1987 Dec;69(9):1328-35. PMID 3440791
- [Background] Cheng T, Chen D, Zhu C, Pan X, Mao X, Guo Y, Zhang X. Fixed- versus mobile-bearing unicondylar knee arthroplasty: are failure modes different? Knee Surg Sports Traumatol Arthrosc. 2013 Nov;21(11):2433-41. doi: 10.1007/s00167-012-2208-y. Epub 2012 Sep 25. PMID 23007412
- [Background] Murray DW, Goodfellow JW, O'Connor JJ. The Oxford medial unicompartmental arthroplasty: a ten-year survival study. J Bone Joint Surg Br. 1998 Nov;80(6):983-9. doi: 10.1302/0301-620x.80b6.8177. PMID 9853489
- [Background] Pandit H, Jenkins C, Gill HS, Smith G, Price AJ, Dodd CA, Murray DW. Unnecessary contraindications for mobile-bearing unicompartmental knee replacement. J Bone Joint Surg Br. 2011 May;93(5):622-8. doi: 10.1302/0301-620X.93B5.26214. PMID 21511927
- [Result] Nam D, Berend ME, Nunley RM, Della Valle CJ, Berend KR, Lombardi AV, Barrack RL. Residual Symptoms and Function After Unicompartmental and Total Knee Arthroplasty: Comparable to Normative Controls? J Arthroplasty. 2016 Oct;31(10):2161-6. doi: 10.1016/j.arth.2016.02.064. Epub 2016 Mar 10. PMID 27067170